CLINICAL TRIAL: NCT04087863
Title: A Multi-center, Open, Single-arm Clinical Trial to Evaluate the Safety and Efficacy of FURESTEM-AD Inj. in Patients With Moderate to Severe Chronic Atopic Dermatitis Who Participated in a Placebo Group in K0102 Clinical Trial: 2nd Extension Study of K0102
Brief Title: Administration for Placebo Group and Evalution the Safety and Efficacy in Atopic Dermatitis Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kang Stem Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: K0103
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Atopic Dermatitis
  Interventions: Other: Not applicable(observational study)

INTERVENTIONS:
Other: Not applicable(observational study) — Not applicable(observational study)

SUMMARY:
A Multi-center, Open, Single-arm Clinical Trial to Evaluate the Safety and Efficacy of FURESTEM-AD inj. in Patients with Moderate to Severe Chronic Atopic Dermatitis Who Participated in a Placebo Group in K0102 Clinical Trial: 2nd Extension Study of K0102

ELIGIBILITY:
Inclusion Criteria:

1. Subject who enrolled K0102 Clinical Trial(parent study) and be assigned to a placebo group
2. Subjects who understand and voluntarily sign an informed consent form

Exclusion Criteria:

1. Subjects with medical history or surgery/procedure history
2. Subjects with diseases at the time of participation in this study (systemic infection, other serious skin disorders, pigmentation or extensive scarring in atopic dermatitis symptom region)
3. Pregnant, breast-feeding women or women who plan to become pregnant during six months after administering the clinical trial medication
4. Subjects who participate in other clinical trial or participated in other clinical trial within 4 weeks
5. In case follow-up is not possible to end of this study period
6. Any other condition which the investigator judges would make patient unsuitable for study participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Moderate to Severe Atopic Dermatitis
Sampling Method: Non-Probability Sample
Enrollment: 99 (Estimated)
Dates: Start 2019-08-29 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety Assessment (Rate of Adverse Event, Number of Participants with Adverse Event) | 5 years

SECONDARY OUTCOMES:
Percentage of subjects whose Eczema Area and Severity Index (EASI) was decreased from baseline by more than 75% at each visit (EASI-75) | 3 years
Percentage of subjects whose Eczema Area and Severity Index (EASI) was decreased from baseline by more than 50% at each visit (EASI-50) | 3 years
Rate of change in EASI from baseline | 3 years
  EASI range is from 0 (clear) to 72 (severe)
Change in EASI from baseline | 3 years
  EASI range is from 0 (clear) to 72 (severe)
Percentage of subjects whose Investigator's Global Assessment (IGA) score at each visit is 0 or 1 | 3 years
Percentage of subjects whose IGA at each visit is 0 or 1, or improved to 2 or higher | 3 years
  IGA score is from 0 (clear) to 5 (severe)
Percentage of subjects whose SCORing Atopic Dermatitis (SCORAD) INDEX was decreased from baseline by more than 50% at each visit (SCORAD-50) | 3 years
Rate of change in SCORAD index from baseline at each visit | 3 years
Change in SCORAD index from baseline at each visit | 3 years
  SCORAD index range is from 0 (clear) to 103 (severe)
Rate of change in Extent, Intensity of lesions and subject symptoms for SCORAD index from baseline at each visit | 3 years
Change in Extent, Intensity of lesions and subject symptoms for SCORAD index from baseline at each visit | 3 years
  SCORAD index range is from 0 (clear) to 103 (severe)
Change in total serum Immunoglobulin E(IgE) from baseline | 3 years
Rate of change in total serum Immunoglobulin E(IgE) from baseline | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided